CLINICAL TRIAL: NCT07394062
Title: A Prospective Observational Study Comparing Chemotherapy Plus Pembrolizumab Versus Nivolumab Plus Ipilimumab With Chemotherapy in Patients With Metastatic Non-Small Cell Lung Cancer and PD-L1 Expression Below 50%
Brief Title: Real-World Comparison of Chemo-Immunotherapy Regimens in Metastatic NSCLC With PD-L1 <50% (ALCG-01)
Acronym: ALCG-01
Status: Recruiting | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Orhun Akdoğan, Medical Oncologist, Gazi University
Other Study IDs: ALCG-01; AEŞH-EK-2025-317 (Other: Ankara Etlik City Hospital Clinical Research Ethics Committee)
Record Dates: First submitted 2026-02-02; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Nonsmall Cell Lung Cancer, Stage IV; Metastatic Nonsmall Cell Lung Cancer
Keywords: NSCLC; Metastatic Lung Cancer; Chemo-Immunotherapy; PD-L1; Progression-Free Survival; Overall Survival; Quality of Life; Patient-Reported Outcomes
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — pembrolizumab; Nivolumab; Ipilimumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chemo + Pembrolizumab: Patients receiving platinum-based chemotherapy combined with pembrolizumab as part of routine care.
  Interventions: Drug: Pembrolizumab
- Nivolumab + Ipilimumab + Chemotherapy: Patients receiving nivolumab plus ipilimumab in combination with platinum-based chemotherapy as part of routine care.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab (1mg/kg)

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab administered as part of routine clinical care in combination with platinum-based chemotherapy, according to standard clinical practice. Treatment selection, dosing, and scheduling are determined by the treating physician and are not protocol-mandated.
  Groups: Chemo + Pembrolizumab
Drug: Nivolumab — Nivolumab administered as part of routine clinical care in combination with ipilimumab and platinum-based chemotherapy, according to standard clinical practice. Treatment selection, dosing, scheduling, and duration are determined by the treating physician and are not protocol-mandated.
  Groups: Nivolumab + Ipilimumab + Chemotherapy
Drug: Ipilimumab (1mg/kg) — Ipilimumab administered as part of routine clinical care in combination with nivolumab and platinum-based chemotherapy, according to standard clinical practice. Treatment selection, dosing, scheduling, and duration are determined by the treating physician and are not protocol-mandated.
  Groups: Nivolumab + Ipilimumab + Chemotherapy

SUMMARY:
Patients with metastatic non-small cell lung cancer (NSCLC) and programmed death-ligand 1 (PD-L1) expression below 50% are commonly treated with different chemo-immunotherapy regimens in routine clinical practice. Although these regimens are widely used, comparative real-world data on survival outcomes and patient-reported quality of life are limited.

This prospective observational study aims to compare two commonly used treatment approaches in patients with metastatic NSCLC and PD-L1 expression <50%: chemotherapy plus pembrolizumab versus nivolumab plus ipilimumab combined with chemotherapy. Patients will receive treatment according to routine clinical decisions made by their treating physicians; no treatment assignment or intervention will be performed as part of the study.

The primary outcomes of the study are progression-free survival and overall survival. In addition, health-related quality of life will be assessed using validated patient-reported outcome questionnaires during routine follow-up.

Exploratory analyses will examine treatment outcomes in relation to selected clinical and patient-related factors, such as biological age, antibiotic exposure, and dietary patterns, in subsets of patients with available data.

The results of this study are expected to provide real-world evidence on survival and quality of life outcomes associated with commonly used chemo-immunotherapy strategies in metastatic NSCLC.

DETAILED DESCRIPTION:
This is a prospective, observational cohort study conducted in patients with metastatic non-small cell lung cancer (NSCLC) and programmed death-ligand 1 (PD-L1) expression below 50% who are treated in routine clinical practice.

Eligible patients will receive systemic treatment according to standard-of-care decisions made by their treating physicians. Two commonly used treatment approaches will be observed: chemotherapy combined with pembrolizumab, and nivolumab plus ipilimumab administered in combination with chemotherapy. No randomization, protocol-driven treatment assignment, or experimental intervention will be performed as part of the study.

The primary objectives of the study are to compare progression-free survival (PFS) and overall survival (OS) between the two treatment approaches. Survival outcomes will be assessed using standard clinical and radiological follow-up data collected during routine care.

Secondary objectives include the evaluation of health-related quality of life and patient-reported outcomes. Quality of life will be assessed using validated questionnaires administered during routine follow-up visits, including global quality of life, functional status, cognitive function, and psychological well-being.

In addition to the primary and secondary objectives, exploratory analyses are planned to investigate the association between treatment outcomes and selected patient-related factors. These include biological age metrics, exposure to antibiotics during treatment, and dietary patterns assessed through patient questionnaires. These analyses will be conducted in subsets of patients with available and complete data for the relevant variables.

As an observational real-world study, missing data are anticipated for some variables, particularly patient-reported and lifestyle-related measures. All analyses will be performed using appropriate statistical methods, and results from exploratory analyses will be interpreted as hypothesis-generating.

This study is designed to provide prospective real-world evidence on the comparative effectiveness and patient-reported outcomes of widely used chemo-immunotherapy regimens in metastatic NSCLC patients with PD-L1 expression below 50%.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Histologically or cytologically confirmed non-small cell lung cancer.
* Metastatic (stage IV) disease at the time of study entry.
* Tumor PD-L1 expression <50%.
* Initiation of first-line systemic treatment with either chemotherapy plus pembrolizumab or nivolumab plus ipilimumab in combination with chemotherapy, according to routine clinical practice.
* Ability to provide informed consent.

Exclusion Criteria:

* Prior systemic therapy for metastatic non-small cell lung cancer.
* Participation in an interventional clinical trial that mandates treatment assignment.
* Presence of another active malignancy requiring systemic treatment.
* Inability to comply with routine clinical follow-up or data collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients with metastatic non-small cell lung cancer and PD-L1 expression below 50% who are receiving standard first-line chemo-immunotherapy regimens in routine clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Up to 18 months
  Progression-free survival, defined as the time from treatment initiation to radiologic disease progression or death from any cause, whichever occurs first, assessed according to routine clinical and radiological evaluations.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 24 months
  Overall survival, defined as the time from treatment initiation to death from any cause.
Health-Related Quality of Life | Up to 18 months
  Health-related quality of life assessed using the EORTC QLQ-C30 questionnaire, including the global health status/quality of life score, administered during routine follow-up.

OTHER OUTCOMES:
Treatment Outcomes According to Antibiotic Exposure | Up to 18 months
  Association between antibiotic exposure during treatment and clinical outcomes, including progression-free survival and overall survival, analyzed in patients with available antibiotic use data.
Treatment Outcomes According to Dietary Patterns | Up to 24 months
  Association between dietary patterns assessed by patient questionnaires and treatment outcomes, including progression-free survival and overall survival, analyzed in a subset of patients with available dietary data.
Treatment Outcomes According to Biological Age | Up to 24 months
  Association between biological age metrics and treatment outcomes, including progression-free survival and overall survival, analyzed in patients with available data.

CONTACTS AND LOCATIONS:
Overall Officials: Ozan Yazıcı, MD, Study Chair — Gazi University
Locations (2):
- Turkey (Türkiye) (2):
  - Ankara Etlik City Hospital, Ankara
  - Gazi University Faculty of Medicine, Department of Medical Oncology, Ankara

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the study involves prospectively collected clinical and patient-reported data obtained as part of routine clinical care, and data sharing was not included in the original study protocol or informed consent. Any data use will be limited to the approved analyses within the study framework.